CLINICAL TRIAL: NCT06661850
Title: A Multi-Center Randomized Clinical Study of the NOCISCAN MR Spectroscopy (MRS) in Patients Treated for Discogenic Low Back Pain
Brief Title: Examination of Nociscan Impact on Discogenic Low Back Pain Surgical Outcomes
Acronym: CLARITY
Status: Recruiting | Type: Observational
Sponsor: Aclarion (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Other Study IDs: Clarity
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Discogenic Low Back Pain
Keywords: MR Spectroscopy; MRI; back pain; Nociscan
MeSH Terms: conditions — Back Pain | interventions — Gene Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Blinded-to-NOCISCAN: NOCISCAN completed pre-operatively. Investigator will not have access to NOCISCAN result.
  Interventions: Procedure: Fusion or TDR determined by investigator.
- Unblinded-to-NOCISCAN: NOCISCAN completed pre-operatively. Investigator will have access to the NOCISCAN result after completing initial treatment plan but before treatment.
  Interventions: Procedure: Fusion or TDR determined by investigator.

INTERVENTIONS:
Procedure: Fusion or TDR determined by investigator. — The surgical treatment will be decided by the treating investigator based on their clinical judgement.

SUMMARY:
This study is looking into how safe and useful NOCISCAN is. NOCISCAN is a software as a Service (SaaS) tool that uses Magnetic Resonance (MR) spectroscopy. Nociscan (instead of 'It') leverages MRS to noninvasively help physicians distinguish between painful and nonpainful discs in the lumbar spine. The randomized controlled trial will compare the blinded and unblinded cohorts and their corresponding surgical outcomes with the Nocigram reports, generated prior to treatment, for each patient."

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a skeletally mature male or female (non-pregnant) aged 18 to 70 years (inclusive);
2. Subject plans to undergo surgical treatment of their discogenic back pain independent of this research protocol;
3. Subject is to be treated with on-label use of FDA-cleared or FDA-approved devices independent of this research protocol;
4. Subject has a diagnosis of discogenic back pain that requires treatment in up to two lumbar levels caused by degenerative disc disease (identified via MRI);
5. Subject has a preoperative Oswestry Disability Questionnaire score ≥35 out of 100 points (35/100);
6. Subject has a VAS back pain score of ≥40mm and that is greater than the worst VAS leg pain score;
7. Subject has failed at least ≥ 6 months of non-operative treatment (for example: physical therapy, bed rest, anti-inflammatory or analgesic medications, chiropractic care, acupuncture, massage therapy or home-directed lumbar exercise programs) OR requires urgent surgical treatment per the investigator;
8. Subject has signed the IRB approved Informed Consent Form; and
9. Subject is psychosocially, mentally and physically able and willing to fully comply with this protocol including adhering to follow-up schedule and requirements and filling out forms.

Exclusion Criteria:

1. Subject has a primary diagnosis of spinal condition other than degenerative disc disease at the involved level (i.e., facet joint pain/SI pain);
2. Subject has had prior lumbar back surgery or intradiscal treatments at any lumbar level (Note: diagnostic provocative or anesthetic discography are not excluded; micro-discectomy, decompression, or laminectomy patients greater than 6 months postop are not excluded);
3. Surgery is planned for more than 2 lumbar levels.
4. Subject has severe spinal canal stenosis as assessed by the Investigator;
5. Subject has a motor strength deficit(s) in lower extremities
6. Subject has a lumbar spine diagnosis, based on radiographic evidence, of clinically relevant lumbar vertebral abnormalities (except Modic end-plate changes, which are not excluded), including:

   * Spondylolisthesis Grade 2 or greater (up to Grade 1 is accepted)
   * Pars fracture, at the involved level
   * Spondylolysis
   * Lumbar scoliosis with a Cobb angle of greater than 15°
   * Evidence of prior fracture or trauma to the L1, L2, L3, L4, or L5 levels in either compression or burst
   * Lumbar kyphosis
7. Subject has radiologic evidence of an uncontained lumbar disc herniation or lumbar disc extrusion.
8. Subject is contraindicated for a standard lumbar MRI exam
9. Women who are currently pregnant (or believe they may be at risk of being or becoming pregnant), or are breast feeding, during the study period when scans will be performed
10. Subject is currently receiving worker's compensation or is involved in in any litigation for personal injury, medical negligence, trauma, or worker's compensation.
11. Subject has a chronic disease (other than degenerative disc disease), chronic pain (other than discogenic low back pain), or psychological dysfunction, which may, in the opinion of the Principal Investigator, compromise a subject's ability to comply with study procedures, and/or may confound data
12. Subject has a BMI > 40

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with back pain potentially caused by lumbar degenerative disc disease. Patients may be symptomatic at one level or two levels. Patients must be indicated for surgical treatment of their discogenic low back pain. Patients must also meet all study inclusion criteria and none of the study exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in back pain on 100mm Visual Analog Scale (VAS) Pain Assessment | Baseline to 12 months
  The primary endpoint is change in back pain as measured on a 100mm VAS Back at 12 months compared to baseline.
  VAS is a measurement instrument that measures the amount of pain that a subject feels ranges across a continuum from none to an extreme amount of pain. Higher scores closer to the extreme pain range indicate worse outcome.

SECONDARY OUTCOMES:
20 mm improvement in back pain on 100mm Visual Analog Scale (VAS) Pain Assessment | From Baseline to each follow up visit (3-Months, 6-Months, 12- Months, and 24 Months)
  VAS is a measurement instrument that measures the amount of pain that a subject feels ranges across a continuum from none to an extreme amount of pain. Higher scores closer to the extreme pain range indicate worse outcome.
20 mm improvement in worst leg pain on a 100mm Visual Analog Scale (VAS) Pain Assessment | From Baseline to each follow up visit (3-Months, 6-Months, 12- Months, and 24 Months)
  VAS is a measurement instrument that measures the amount of pain that a subject feels ranges across a continuum from none to an extreme amount of pain. Higher scores closer to the extreme pain range indicate worse outcome.
Patient reported treatment satisfaction survey | Each follow up visit (3-Months, 6-Months, 12- Months, and 24 Months)
  Patient Satisfaction survey is a self-reported questionnaire to measure the subject's satisfaction of the treatment under the protocol.
Patient-Reported Outcome Measurement Information System (PROMIS) 29 score | Each follow up visit (3-Months, 6-Months, 12- Months, and 24 Months)
  The PROMIS-29 v2. 0 profile assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain.
Cumulative proportion of responders (CPRA) for 15 point Oswestry Disability Index (ODI) change (out of 100) | From Baseline to each follow up visit (3-Months, 6-Months, 12- Months, and 24 Months)
  The Oswestry Disability Index (ODI) is a 10-item questionnaire that scores disability on a percentile scale from 0-100%. The ODI score is interpreted as follows:
  0-20%: Minimal disability 20-40%: Moderate disability 40-60%: Severe disability 60-80%: Crippling effects 80-100%: Completely disabled and bedbound
Absence of Secondary surgical intervention | From Baseline through study completion, 24-Months
  Secondary surgical interventions may include revision, reoperation, removal or supplemental fixation at any level in the lumbar spine.
Correlation of preoperative NOCISCAN Biomarkers with preoperative Visual Analog Scale (VAS) Pain Assessment Scores | From Baseline through study completion, 24-Months
  VAS is a measurement instrument that measures the amount of pain that a subject feels ranges across a continuum from none to an extreme amount of pain. Higher scores closer to the extreme pain range indicate worse outcome.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Scripps Health, La Jolla, California
  - USC Keck Medical Center, Los Angeles, California
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Advocate Aurora Research Institute, Park Ridge, Illinois
  - Texas Back Institute, Plano, Texas

REFERENCES:
- See also: Related Info — https://aclarion.com/